CLINICAL TRIAL: NCT06198946
Title: External Diaphragm Pacing Therapy and Correlation Analysis of Trunk Balance and Respiratory Function in Stroke Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The first phase of the research has been completed
Sponsor: Zhang liqiong (Other)
Responsible Party: Sponsor-Investigator, Zhang liqiong, resident physician, The First Affiliated Hospital of Anhui Medical University
Organization: The First Affiliated Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Zliqiong
Record Dates: First submitted 2023-12-13; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Stroke; Respiratory Function
Keywords: External diaphragm pacing; Respiratory function; Diaphragm function; Stroke
MeSH Terms: conditions — Stroke; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Provide participants with routine rehabilitation treatment
  Interventions: Other: Routine rehabilitation treatment
- observation group (Other): Participants received EDP treatment on the basis of conventional rehabilitation treatment
  Interventions: Device: External diaphragm pacing（EDP）; Other: Routine rehabilitation treatment

INTERVENTIONS:
Device: External diaphragm pacing（EDP） — After the skin is disinfected, place the small electrode pads on the lower 1/3 of the outer edges of the sternocleidomastoid muscles on the left and right sides, and place the large electrodes on the surface of the pectoralis major muscles on both sides, and fix them with medical tape. Adjust the pacing according to the patient's tolerance. Frequency and stimulation intensity, each treatment time is 20 minutes, treatment is once a day, 5 days a week, and the treatment course is 4 weeks.
  Arms: observation group
Other: Routine rehabilitation treatment — Participants received comprehensive rehabilitation treatments such as muscle strength training, hemiplegic limb comprehensive training, balance function training, limb neuromuscular electrical stimulation, acupuncture and other comprehensive rehabilitation treatments. Each project was 30 minutes/time, once a day, 5 days a week, and the treatment course was 4 weeks.comprehensive rehabilitation treatments, each item is 30 minutes/time, once a day, 5 days a week, and the treatment course is 4 weeks.

SUMMARY:
The goal of this study is to observe the enhancement of trunk balance ability, pulmonary function, and diaphragm function in stroke patients after treatment of external diaphragm pacing（EDP）, and analyze the potential correlation between trunk balance ability and respiratory function metrics. The main questions it aims to answer are:

* What is the effect of EDP treatment on trunk balance and respiratory function in stroke patients?
* Is there a correlation between trunk balance ability and respiratory function?

Participants admitted to the Department of Rehabilitation Medicine at the First Affiliated Hospital of Anhui Medical University were randomly divided into an observation group and a control group：

* The control group received conventional rehabilitation therapy for 4 weeks.
* The observation group received EDP treatment in addition to conventional rehabilitation therapy for 4 weeks.

DETAILED DESCRIPTION:
Objective：To observe the enhancement of trunk balance ability, pulmonary function, and diaphragm function in stroke patients after treatment of external diaphragm pacing（EDP）, and analyze the potential correlation between trunk balance ability and respiratory function metrics.

Methods：Thirty stroke patients admitted to the Department of Rehabilitation Medicine at the First Affiliated Hospital of Anhui Medical University from January 2023 to August 2023 were selected. They were randomly divided into an observation group (n=15) and a control group (n=15). The control group received conventional rehabilitation therapy, while the observation group received EDP treatment in addition to conventional rehabilitation therapy for 4 weeks. Independent sample t-tests and rank-sum tests were used to compare the Modified Trunk Impairment Scale (mTIS) scores, Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1), FEV1/FVC change in percentage of Vital Capacity from sitting to supine position (ΔVC), diaphragmatic excursion of quiet breath(DE-QB), diaphragmatic excursion of deep breath (DE-DB), and Thickening Fraction (TF) between the two groups of patients. Pearson correlation analysis was employed to explore the correlations among these indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for stroke for the first time;
* Patients whose disease duration is within 6 months, have received specialist and standardized treatment, and have stable vital signs;
* Patients are informed of this study, voluntarily accept rehabilitation treatment, and sign an informed consent form;
* Patients who have no chronic breathing before and after stroke History of systemic and circulatory diseases.
* The patient can maintain the starting posture evaluated by the mTIS scale for 10 seconds. The standard for the starting posture is: sitting on the edge of the bed without any support for the back and arms, with the thighs in full contact with the bed surface, and with the feet flat and the same width as the hips. On the ground, bend your knees 90° and place your arms on your thighs .

Exclusion Criteria:

* Those who are complicated by severe heart, lung and other organ dysfunction diseases, such as pulmonary embolism, pacemaker placement, etc.;
* Those who are complicated by severe cognitive impairment and abnormal hearing and understanding;
* There are other reasons why electrical stimulation treatment is not suitable, Such as sudden unstable vital signs, malignant tumors, combined with mental illness, etc.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity(FVC) | Day 1 (before starting treatment) and 4 weeks later
  It is used to assess Respiratory function.FVC was evaluated using an exercise cardiopulmonary testing system (Nanjing Hanya Smax58ce).
Forced Expiratory Volume in 1 second (FEV1) | Day 1 (before starting treatment) and 4 weeks later
  It is used to assess Respiratory function.FEV1 was evaluated using an exercise cardiopulmonary testing system (Nanjing Hanya Smax58ce).
Forced expiratory volume in 1 second as a percentage of forced vital capacity(FEV1/FVC) | Day 1 (before starting treatment) and 4 weeks later
  It is used to assess Respiratory function.FEV1/FVC(%) was evaluated using an exercise cardiopulmonary testing system (Nanjing Hanya Smax58ce).
diaphragmatic excursion of deep breath(DE-DB） | Day 1 (before starting treatment) and 4 weeks later
  It is used to assess Respiratory function.DE-DB was evaluated using Sonoson portable color ultrasound (M-Turbo).
Thickening Fraction(TF) | Day 1 (before starting treatment) and 4 weeks later
  It is used to assess Respiratory function.TF was evaluated using Sonoson portable color ultrasound (M-Turbo).
diaphragmatic excursion of quiet breath(ED-QB) | Day 1 (before starting treatment) and 4 weeks later
  It is used to assess Respiratory function.DE-QB was evaluated using Sonoson portable color ultrasound (M-Turbo).
the Modified Trunk Impairment Scale (mTIS) | Day 1 (before starting treatment) and 4 weeks later
  It is used to assess trunk balance ability and includes the dynamic seated balance subscale (10 points) and the coordination subscale (6 points), with a total score of 16 points.

CONTACTS AND LOCATIONS:
Overall Officials: Liqiong Zhang, Study Chair — Anhui Medical University
Locations (1):
- Zhangliqiong, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-09-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT06198946/Prot_000.pdf
  • Informed Consent Form (2022-09-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT06198946/ICF_001.pdf